CLINICAL TRIAL: NCT00626496
Title: Genetic Epidemiology of Lymphoproliferative Disorders
Brief Title: Family Study of Lymphoproliferative Disorders
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan Slager, Professor, Mayo Clinic
Other Study IDs: 489-04; U01CA118444 (NIH); R01CA235026 (NIH); NCI-2021-14099 (Registry Identifier: CTRP); LS0587 (Other: Mayo Clinic)
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Monoclonal B-Cell Lymphocytosis; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Multiple Myeloma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect blood samples from patients and their relatives for DNA and cytogenetic studies. A one time blood draw of 50 cc will be done.
Oversight: Data Monitoring Committee: No

SUMMARY:
Blood and lymph node cancers can begin in either the lymphatic tissues (as in the case of lymphoma) or in the bone marrow (as with leukemia and myeloma), and they all are involved with the uncontrolled growth of white blood cells. There are many subtypes of these cancers, e.g., chronic lymphocytic leukemia and non-Hodgkin lymphoma. Since there is evidence that these cancers cluster in families, this study aims to understand how genetics and environmental exposures contribute to the development of these cancers.

ELIGIBILITY:
At least 2 living, blood related relatives, affected with a lymphoproliferative disorder.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over the age of 18 who have a family history of a blood or lymph node disorder.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2004-04-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of blood or lymphoma | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slager, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Sellick GS, Goldin LR, Wild RW, Slager SL, Ressenti L, Strom SS, Dyer MJ, Mauro FR, Marti GE, Fuller S, Lyttelton M, Kipps TJ, Keating MJ, Call TG, Catovsky D, Caporaso N, Houlston RS. A high-density SNP genome-wide linkage search of 206 families identifies susceptibility loci for chronic lymphocytic leukemia. Blood. 2007 Nov 1;110(9):3326-33. doi: 10.1182/blood-2007-05-091561. Epub 2007 Aug 8. PMID 17687107
- [Result] Slager SL, Kay NE, Fredericksen ZS, Wang AH, Liebow M, Cunningham JM, Vachon CM, Call TG, Cerhan JR. Susceptibility genes and B-chronic lymphocytic leukaemia. Br J Haematol. 2007 Dec;139(5):762-71. doi: 10.1111/j.1365-2141.2007.06872.x. PMID 18021089
- [Result] Caporaso N, Goldin L, Plass C, Calin G, Marti G, Bauer S, Raveche E, McMaster ML, Ng D, Landgren O, Slager S. Chronic lymphocytic leukaemia genetics overview. Br J Haematol. 2007 Dec;139(5):630-4. doi: 10.1111/j.1365-2141.2007.06846.x. PMID 18021078
- [Result] Goldin LR, Slager SL. Familial CLL: genes and environment. Hematology Am Soc Hematol Educ Program. 2007:339-45. doi: 10.1182/asheducation-2007.1.339. PMID 18024649
- [Result] Slager SL, Kay NE. Familial chronic lymphocytic leukemia: what does it mean to me? Clin Lymphoma Myeloma. 2009;9 Suppl 3(Suppl 3):S194-7. doi: 10.3816/CLM.2009.s.011. PMID 19778840
- [Result] Slager SL, Goldin LR, Strom SS, Lanasa MC, Spector LG, Rassenti L, Leis JF, Camp NJ, Kay NE, Vachon CM, Glenn M, Weinberg JB, Rabe KG, Cunningham JM, Achenbach SJ, Hanson CA, Marti GE, Call TG, Caporaso NE, Cerhan JR. Genetic susceptibility variants for chronic lymphocytic leukemia. Cancer Epidemiol Biomarkers Prev. 2010 Apr;19(4):1098-102. doi: 10.1158/1055-9965.EPI-09-1217. Epub 2010 Mar 23. PMID 20332261
- [Result] Conde L, Halperin E, Akers NK, Brown KM, Smedby KE, Rothman N, Nieters A, Slager SL, Brooks-Wilson A, Agana L, Riby J, Liu J, Adami HO, Darabi H, Hjalgrim H, Low HQ, Humphreys K, Melbye M, Chang ET, Glimelius B, Cozen W, Davis S, Hartge P, Morton LM, Schenk M, Wang SS, Armstrong B, Kricker A, Milliken S, Purdue MP, Vajdic CM, Boyle P, Lan Q, Zahm SH, Zhang Y, Zheng T, Becker N, Benavente Y, Boffetta P, Brennan P, Butterbach K, Cocco P, Foretova L, Maynadie M, de Sanjose S, Staines A, Spinelli JJ, Achenbach SJ, Call TG, Camp NJ, Glenn M, Caporaso NE, Cerhan JR, Cunningham JM, Goldin LR, Hanson CA, Kay NE, Lanasa MC, Leis JF, Marti GE, Rabe KG, Rassenti LZ, Spector LG, Strom SS, Vachon CM, Weinberg JB, Holly EA, Chanock S, Smith MT, Bracci PM, Skibola CF. Genome-wide association study of follicular lymphoma identifies a risk locus at 6p21.32. Nat Genet. 2010 Aug;42(8):661-4. doi: 10.1038/ng.626. Epub 2010 Jul 18. PMID 20639881
- [Result] Goldin LR, Slager SL, Caporaso NE. Familial chronic lymphocytic leukemia. Curr Opin Hematol. 2010 Jul;17(4):350-5. doi: 10.1097/MOH.0b013e328338cd99. PMID 20389242
- [Result] Goldin LR, Lanasa MC, Slager SL, Cerhan JR, Vachon CM, Strom SS, Camp NJ, Spector LG, Leis JF, Morrison VA, Glenn M, Rabe KG, Achenbach SJ, Algood SD, Abbasi F, Fontaine L, Yau M, Rassenti LZ, Kay NE, Call TG, Hanson CA, Weinberg JB, Marti GE, Caporaso NE. Common occurrence of monoclonal B-cell lymphocytosis among members of high-risk CLL families. Br J Haematol. 2010 Oct;151(2):152-8. doi: 10.1111/j.1365-2141.2010.08339.x. Epub 2010 Aug 25. PMID 20738309
- [Result] Slager SL, Rabe KG, Achenbach SJ, Vachon CM, Goldin LR, Strom SS, Lanasa MC, Spector LG, Rassenti LZ, Leis JF, Camp NJ, Glenn M, Kay NE, Cunningham JM, Hanson CA, Marti GE, Weinberg JB, Morrison VA, Link BK, Call TG, Caporaso NE, Cerhan JR. Genome-wide association study identifies a novel susceptibility locus at 6p21.3 among familial CLL. Blood. 2011 Feb 10;117(6):1911-6. doi: 10.1182/blood-2010-09-308205. Epub 2010 Dec 3. PMID 21131588
- [Result] Lanasa MC, Allgood SD, Slager SL, Dave SS, Love C, Marti GE, Kay NE, Hanson CA, Rabe KG, Achenbach SJ, Goldin LR, Camp NJ, Goodman BK, Vachon CM, Spector LG, Rassenti LZ, Leis JF, Gockerman JP, Strom SS, Call TG, Glenn M, Cerhan JR, Levesque MC, Weinberg JB, Caporaso NE. Immunophenotypic and gene expression analysis of monoclonal B-cell lymphocytosis shows biologic characteristics associated with good prognosis CLL. Leukemia. 2011 Sep;25(9):1459-66. doi: 10.1038/leu.2011.117. Epub 2011 May 27. PMID 21617698
- [Result] Campa D, Butterbach K, Slager SL, Skibola CF, de Sanjose S, Benavente Y, Becker N, Foretova L, Maynadie M, Cocco P, Staines A, Kaaks R, Boffetta P, Brennan P, Conde L, Bracci PM, Caporaso NE, Strom SS, Camp NJ, Cerhan JR; GEC Consortium; Canzian F, Nieters A. A comprehensive study of polymorphisms in the ABCB1, ABCC2, ABCG2, NR1I2 genes and lymphoma risk. Int J Cancer. 2012 Aug 15;131(4):803-12. doi: 10.1002/ijc.26436. Epub 2011 Nov 28. PMID 21918980
- [Result] Slager SL, Skibola CF, Di Bernardo MC, Conde L, Broderick P, McDonnell SK, Goldin LR, Croft N, Holroyd A, Harris S, Riby J, Serie DJ, Kay NE, Call TG, Bracci PM, Halperin E, Lanasa MC, Cunningham JM, Leis JF, Morrison VA, Spector LG, Vachon CM, Shanafelt TD, Strom SS, Camp NJ, Weinberg JB, Matutes E, Caporaso NE, Wade R, Dyer MJ, Dearden C, Cerhan JR, Catovsky D, Houlston RS. Common variation at 6p21.31 (BAK1) influences the risk of chronic lymphocytic leukemia. Blood. 2012 Jul 26;120(4):843-6. doi: 10.1182/blood-2012-03-413591. Epub 2012 Jun 13. PMID 22700719
- [Result] Coombs CC, Rassenti LZ, Falchi L, Slager SL, Strom SS, Ferrajoli A, Weinberg JB, Kipps TJ, Lanasa MC. Single nucleotide polymorphisms and inherited risk of chronic lymphocytic leukemia among African Americans. Blood. 2012 Aug 23;120(8):1687-90. doi: 10.1182/blood-2012-02-408799. Epub 2012 Jun 28. PMID 22745306
- [Result] Slager SL, Camp NJ, Conde L, Shanafelt TD, Achenbach SJ, Rabe KG, Kay NE, Novak AJ, Call TG, Bracci PM, Sille FM, Sanchez S, Akers NK, Cunningham JM, Serie DJ, McDonnell SK, Leis JF, Wang AH, Weinberg JB, Glenn M, Link B, Vachon CM, Lanasa MC, Skibola CF, Cerhan JR. Common variants within 6p21.31 locus are associated with chronic lymphocytic leukaemia and, potentially, other non-Hodgkin lymphoma subtypes. Br J Haematol. 2012 Dec;159(5):572-6. doi: 10.1111/bjh.12070. Epub 2012 Oct 1. PMID 23025533
- [Result] Hebbring SJ, Slager SL, Epperla N, Mazza JJ, Ye Z, Zhou Z, Achenbach SJ, Vasco DA, Call TG, Rabe KG, Kay NE, Caporaso NE, Lanasa MC, Camp NJ, Strom SS, Goldin LR, Cerhan JR, Brilliant MH, Schrodi SJ. Genetic evidence of PTPN22 effects on chronic lymphocytic leukemia. Blood. 2013 Jan 3;121(1):237-8. doi: 10.1182/blood-2012-08-450221. No abstract available. PMID 23287625
- [Result] Slager SL, Achenbach SJ, Asmann YW, Camp NJ, Rabe KG, Goldin LR, Call TG, Shanafelt TD, Kay NE, Cunningham JM, Wang AH, Weinberg JB, Norman AD, Link BK, Leis JF, Vachon CM, Lanasa MC, Caporaso NE, Novak AJ, Cerhan JR. Mapping of the IRF8 gene identifies a 3'UTR variant associated with risk of chronic lymphocytic leukemia but not other common non-Hodgkin lymphoma subtypes. Cancer Epidemiol Biomarkers Prev. 2013 Mar;22(3):461-6. doi: 10.1158/1055-9965.EPI-12-1217. Epub 2013 Jan 10. PMID 23307532
- [Result] Berndt SI, Skibola CF, Joseph V, Camp NJ, Nieters A, Wang Z, Cozen W, Monnereau A, Wang SS, Kelly RS, Lan Q, Teras LR, Chatterjee N, Chung CC, Yeager M, Brooks-Wilson AR, Hartge P, Purdue MP, Birmann BM, Armstrong BK, Cocco P, Zhang Y, Severi G, Zeleniuch-Jacquotte A, Lawrence C, Burdette L, Yuenger J, Hutchinson A, Jacobs KB, Call TG, Shanafelt TD, Novak AJ, Kay NE, Liebow M, Wang AH, Smedby KE, Adami HO, Melbye M, Glimelius B, Chang ET, Glenn M, Curtin K, Cannon-Albright LA, Jones B, Diver WR, Link BK, Weiner GJ, Conde L, Bracci PM, Riby J, Holly EA, Smith MT, Jackson RD, Tinker LF, Benavente Y, Becker N, Boffetta P, Brennan P, Foretova L, Maynadie M, McKay J, Staines A, Rabe KG, Achenbach SJ, Vachon CM, Goldin LR, Strom SS, Lanasa MC, Spector LG, Leis JF, Cunningham JM, Weinberg JB, Morrison VA, Caporaso NE, Norman AD, Linet MS, De Roos AJ, Morton LM, Severson RK, Riboli E, Vineis P, Kaaks R, Trichopoulos D, Masala G, Weiderpass E, Chirlaque MD, Vermeulen RC, Travis RC, Giles GG, Albanes D, Virtamo J, Weinstein S, Clavel J, Zheng T, Holford TR, Offit K, Zelenetz A, Klein RJ, Spinelli JJ, Bertrand KA, Laden F, Giovannucci E, Kraft P, Kricker A, Turner J, Vajdic CM, Ennas MG, Ferri GM, Miligi L, Liang L, Sampson J, Crouch S, Park JH, North KE, Cox A, Snowden JA, Wright J, Carracedo A, Lopez-Otin C, Bea S, Salaverria I, Martin-Garcia D, Campo E, Fraumeni JF Jr, de Sanjose S, Hjalgrim H, Cerhan JR, Chanock SJ, Rothman N, Slager SL. Genome-wide association study identifies multiple risk loci for chronic lymphocytic leukemia. Nat Genet. 2013 Aug;45(8):868-76. doi: 10.1038/ng.2652. Epub 2013 Jun 16. PMID 23770605